CLINICAL TRIAL: NCT02448524
Title: A Prospective, Single-blinded, Multi-center, Randomized, Controlled, Registered Clinical Trial on the Efficacy and Safety of Sirolimus-eluting Stent (MiStent® System) in the Treatment of Patients With Coronary Heart Disease
Brief Title: Clinical Trial on the Efficacy and Safety of Sirolimus-Eluting Stent (MiStent® System)
Acronym: DESSOLVE-C
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Micell Technologies (Industry)
Collaborators: Hefei Life Science Medical Instruments Co. Ltd. (Unknown); Giant Med-Pharma Services Inc. (Industry); CCRF Consulting Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MiStent01
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Coronary Heart Disease
Keywords: Treatment; patients; primary in situ CHD (de novo) lesions
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MiStentTM (Experimental): MiStentTM coronary drug eluting stent (MiStent SES) consists of four parts: a bare-metal stent (BMS), a delivery system, resorbable polymer coating and anti-proliferative drug (sirolimus).
  Interventions: Device: MiStent
- TIVOLI (Active Comparator): TIVOLI stent is a mature and fully degradable coating on a cobalt-chromium alloy drug-eluting stent on the market, findings of four years fully demonstrated the efficacy and safety of sirolimus-coated TIVOLI stent.
  Interventions: Device: TIVOLI

INTERVENTIONS:
Device: MiStent — Primary in situ coronary artery disease patients (all patients enrolled with a maximum of two target lesions in different blood vessels and maximum of 2 stents per lesion. Lesions with reference diameter of 2.5mm-3.5mm (by visual measurement) and with length ≤40mm (by visual measurement).
  Arms: MiStentTM
Device: TIVOLI — Primary in situ coronary artery disease patients (all patients enrolled with a maximum of two target lesions in different blood vessels and maximum of 2 stents per lesion. Lesions with reference diameter of 2.5mm-3.5mm (by visual measurement) and with length ≤40mm (by visual measurement).
  Arms: TIVOLI

SUMMARY:
* To evaluate the safety and efficacy of MiStent drug (sirolimus)-eluting stent system in the treatment of coronary heart disease (CHD) in patients with primary in situ CHD (de novo);
* To evaluate operating performance of the MiStent drug (sirolimus)-eluting coronary stent system.

DETAILED DESCRIPTION:
* The study will enroll a total of 428 cases of primary in situ coronary artery disease patients (all patients enrolled with a maximum of two target lesions in different blood vessels and maximum of 2 stents per lesion. If more stents are needed for implantation, stents with the same brand are required, and mixing brands is not allowed for each patient except for salvage with implantation of other brand of stents.)
* Lesions with reference diameter of 2.5mm-3.5mm (by visual measurement) and with length ≤40mm (by visual measurement) will be selected, subjects meeting the inclusion and exclusion criteria and who agree to participate will be enrolled.
* Prospective, single-blinded, multi-center, randomized, controlled clinical trial;
* Patients with in situ primary CHD;
* Clinical sites: up to 18; patients will be enrolled in a 1:1 ratio (i.e., 214 cases enrolled into each group, the MiStent stent group and TIVOLI stent group);
* Clinical follow-up time points: 1 month, 6 months, 9 months, 12 months and yearly at 2-5 years post index procedure;
* Angiographic follow-up at 9 months post index procedure; in-stent late lumen loss measured by quantitative coronary angiography (QCA) will be used as the primary efficacy endpoint for product evaluation;
* In this trial, the collection, collation, statistical analysis and adjudication of all relevant clinical and angiographic data will be conducted by an independent coronary angiography core laboratory (CCRF Medical Technology Co., Ltd.), data management and statistical center, clinical events committee and clinical audit agency. All patients will be followed up for 5 years (by telephone or outpatient form), and the incidence of adverse events will be recorded to allow a more accurate and reliable evaluation of the long-term safety of the MiStentTM drug (sirolimus) eluting coronary stent system.

ELIGIBILITY:
Inclusion Criteria:

* Stable and unstable angina pectoris (AP), old myocardial infarction (OMI), or confirmed evidence of myocardial ischemia;
* Primary in situ coronary artery lesions (up to two target lesions and up to 2 stents per lesion);
* Visual target lesion length ≤40mm;
* Visual reference vessel diameter of 2.5-3.5mm;
* Visual diameter stenosis ≥70%;
* Patients with indications for coronary artery bypass surgery (CABG);
* Subjects participate voluntarily and signed an informed consent willing to accept angiographic and clinical follow-up.

Exclusion Criteria:

* Acute myocardial infarction (AMI) occurred within 7 days prior to the procedure; post-MI complicated with elevated levels of cardiac enzymes (CK-MB, cTNT / I);
* CTO (TIMI-0) lesions, left main lesions, ostial lesions,bypass graft lesions, bifurcation lesions (lateral side branch reference vessel diameter≥2.5mm), restenosis in-stent and three-vessel disease that need to be treated;
* Severe calcified lesions for which balloon pre-dilation is expected to be unsuccessful;
* Tortuous lesions that render stent crossing difficult;
* NYHA class≥III or left ventricular ejection fraction <40%;
* Implantation of other stents in the past year;
* Pregnant or breast-feeding patients or patients planning to get pregnant within the following year;
* Subjects with bleeding tendency or coagulation disorder or PCI contraindications and / or anticoagulant therapy contraindications or who have not tolerated dual antiplatelet treatment within a year to date;
* Presence of other diseases (such as cancer, malignancies, congestive heart failure, organ transplantation or candidate for it) or history of substance abuse (alcohol, cocaine, heroin, etc.), poor protocol compliance or life expectancy of less than 1 year;
* Allergic to one of following: aspirin, heparin, clopidogrel, sirolimus (rapamycin), PLGA polymers, contrast agents and metal;
* Severe liver and kidney dysfunction (ALT or AST level 3 times greater than the upper limit of normal; eGFR <30ml/min);
* Patients participating in any other clinical trial and who have not completed follow-up to the primary endpoint;
* Study subjects with poor compliance judged by investigators, with poor possibility to complete study in accordance with requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
In-stent late lumen loss (LLL) | 9 months post index procedure
  Late lumen loss is the difference in millimeters between the diameter of a stented segment post-procedure compared with the follow-up angiogram at nine months

SECONDARY OUTCOMES:
Success rate of stent implantation (including device success, lesion success and clinical success); | Baseline
Restenosis rate in-stent, at proximal and distal edges of the stent and in-lesion segments; and late lumen loss and percent diameter stenosis in lesion segments | 9 months
Device-related clinical cardiovascular composite endpoints post index procedure, including cardiac death, target vessel myocardial infarction and clinical symptoms driven target lesion revascularization (i.e., target lesion failure [TLF]) | 30 days, 6 months, 12 months, and 2-5 years
Patient-related clinical cardiovascular composite endpoints post index procedure, including all-cause death (cardiac and non-cardiac), nonfatal myocardial infarction and any revascularization | 30 days, 6 months, 12 months and 2-5 years
Incidence of ARC-defined stent thrombosis (definite, probable, possible stent thrombosis at early, late and very late periods) | 30 days, 6 months, 12 months and 2-5 years
Drug-related adverse events of dual antiplatelet therapy (DAPT) post index procedure. | 30 days, 6 months, 12 months and 2-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, MD, Principal Investigator — The General Hospital of Shenyang Military Region
Locations (16):
- China (16):
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Baotou University, Baotou, Inner Mongolia
  - Inner Mongolia People'S Hospital, Hohhot, Inner Mongolia
  - The First Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of Xi'An Jiaotong University, Xi'an, Shaanxi
  - Sir Run Run Shaw Hospital School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The General Hospital of Shenyang Military Region, Area of Shenyang
  - Fu Wai Hospital, National Center for Cardiovascular Disease, Beijing
  - The First Hospital of Jilin University, Changchun
  - The Second Xiangya Hospital of Central South University, Changsha
  - The First Hospital of Lanzhou University, Lanzhou
  - Shanghai Ninth People's Hospital, Shanghai
  - West China Hospital, Sichuan University, Sichuan
  - The Second Hospital of Shanxi Medical University, Taiyuan
  - TEDA International Cardiovascular Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No